CLINICAL TRIAL: NCT01520051
Title: The Efficacy of Mepolizumab Treatment on Rhinovirus Induced Asthma Exacerbations
Brief Title: Mepolizumab Treatment for Rhinovirus-induced Asthma Exacerbations
Acronym: MATERIAL
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: The Netherlands Asthma Foundation (Other); GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Suzanne Bal, Postdoc, investigator of the study, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: MATERIAL
Record Dates: First submitted 2012-01-25; First posted 2012-01-27 (Estimated); Last update posted 2012-02-07 (Estimated); Status verified 2012-02

CONDITIONS: Asthma; Viral Infection
Keywords: Asthma; Viral; Infection; Inflammation; Mepolizumab; Eosinophilia
MeSH Terms: conditions — Asthma; Virus Diseases; Infections; Inflammation; Eosinophilia | interventions — mepolizumab

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mepolizumab (Experimental)
  Interventions: Drug: Mepolizumab
- Saline (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mepolizumab — 3 monthly intravenous infusions of 750 mg
  Other Names: Mepolizumab, SB240563
  Arms: Mepolizumab
Drug: Placebo — 3 monthly intravenous infusions with saline
  Arms: Saline

SUMMARY:
Asthma is a chronic inflammatory disorder of the airways characterized by lower respiratory tract (LRT) symptoms such as wheeze, cough and airway obstruction. Patients with asthma frequently suffer from exacerbations, which can be triggered by allergens and, in particular, viral respiratory infections. It has recently been shown that mepolizumab, a humanized monoclonal antibody that neutralizes interleukin(IL)-5, markedly reduces the exacerbation rate in asthma patients with eosinophilic airway inflammation. Previous studies have indicated that in a mixed population (eosinophilic and non eosinophilic) of mild asthma patients, mepolizumab did not have an impact on lung function and asthma symptom scores upon allergen provocation, although it did on markers such as sputum and blood eosinophils. Together, these observations led to the hypothesis that mepolizumab treatment reduces the exacerbation rate by limiting virus-induced asthma exacerbations.

The investigators hypothesize that neutralization of IL-5 during virus infection in patients with allergic asthma:

1. Reduces virus-induced bronchial inflammation
2. Attenuates virus-induced asthma symptoms, airflow limitation and bronchial hyperresponsiveness.
3. Enhances cellular immune responses to the virus.

The aims of this study are to:

1. To investigate whether IL-5 neutralization reduces the inflammatory response to viral airway infections in allergic asthma patients
2. To investigate whether IL-5 neutralization prevents or reduces asthma symptoms during virus-induced asthma exacerbations
3. To investigate whether IL-5 neutralization affects the cellular immune response to viral airway infections in allergic asthma patients

DETAILED DESCRIPTION:
Mild allergic asthma subjects receive three times an infusion containing 750 mg of mepolizumab. Two weeks after the third infusion, subjects will be experimentally infected with RV16. One day before and six days after infection a bronchoscopy will be performed to collect bronchoalveolar lavage fluid and bronchial brushes. Blood will be collected at each infusion and each bronchoscopy and at least 6 weeks after infection. Lung function will be evaluated throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 - 50 years
* History of episodic chest tightness and wheezing
* Intermittent or mild persistent asthma according to the criteria by the Global Initiative for Asthma
* Non-smoking or stopped smoking more than 12 months ago and ≤ 5 pack years (PY)
* Clinically stable, no history of exacerbations within the last 6 weeks prior to the study
* Steroid-naïve or those patients who are currently not on corticosteroids and have not taken any corticosteroids by any dosing-routes within 2 weeks prior to the study. Occasional usage of inhaled short-acting beta2-agonists as rescue medication is allowed, prior and during the study
* Baseline FEV1 > 80% of predicted
* Airway hyperresponsiveness, indicated by a positive acetyl-ß-methylcholine bromide (MeBr) challenge with PC20 < 9.8 mg/ml
* Positive skin prick test (SPT) to one or more of the 12 common aeroallergen extracts, defined as a wheal with an average diameter of > 3mm
* No other clinically significant abnormality on medical history and clinical examination

Exclusion Criteria:

* Presence of antibodies directed against RV16 in serum (titer > 4), measured at visit 1
* History of clinical significant hypotensive episodes or symptoms of fainting, dizziness, or light-headedness
* Women who are pregnant, lactating or who have a positive urine pregnancy test at visit 1
* Chronic use of any other medication for treatment of lung disease other than short-acting beta2-agonists
* Participation in any clinical investigational drug treatment protocol within the preceding 3 months
* Ongoing use of tobacco products of any kind or previous usage with ≥ 6 total PY
* Concomitant disease or condition which could interfere with the conduct of the study, or for which the treatment might interfere with the conduct of the study, or which would, in the opinion of the investigator, pose an unacceptable risk to the patient
* People with young children (< 2 years)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2012-01; Primary Completion 2013-12 (Estimated); Study Completion 2014-03 (Estimated)

PRIMARY OUTCOMES:
FEV1 | 1 day prior and 6 days after RV16 challenge
  Change in pre-bronchodilator FEV1 between day 70 and day 77, i.e. 1 day prior and 6 days after RV16 challenge.
Questionnaire to score asthma and common cold complaints | During 14 days following viral infection

SECONDARY OUTCOMES:
Viral load | Day 6 after viral infection
  Viral load in nasal swab and bronchial brushes
Sputum eosinophils | Before and after mepolizumab infusion
  Change in sputum eosinophils
Cell influx in bronchoalveolar lavage fluid | 6 days after viral infection
  Influx of neutrophils, eosinophils, macrophages, monocytes, T en B lymphocytes into the lungs
Pro-inflammatory cytokines in bronchoalveolar lavage fluid | 6 days after viral infection
  Measurement of IL-6, IL-8 and IFN-y in bronchoaveolar lavage fluid
Antibody production | 6 weeks after infection
  Anti RV-16 antibodies are measured in serum

CONTACTS AND LOCATIONS:
Overall Officials: René Lutter, PhD, Principal Investigator — Academic Medical Center, Respiratory Medicine; Elisabeth H Bel, MD, PhD, Study Director — Academic Medical Center, Respiratory Medicine; Peter J Sterk, PhD, Study Director — Academic Medical Center, Respiratory Medicine
Locations (1):
- Academic Medical Center, Amsterdam, Netherlands

REFERENCES:
- [Background] Nair P, Pizzichini MM, Kjarsgaard M, Inman MD, Efthimiadis A, Pizzichini E, Hargreave FE, O'Byrne PM. Mepolizumab for prednisone-dependent asthma with sputum eosinophilia. N Engl J Med. 2009 Mar 5;360(10):985-93. doi: 10.1056/NEJMoa0805435. PMID 19264687
- [Background] Haldar P, Brightling CE, Hargadon B, Gupta S, Monteiro W, Sousa A, Marshall RP, Bradding P, Green RH, Wardlaw AJ, Pavord ID. Mepolizumab and exacerbations of refractory eosinophilic asthma. N Engl J Med. 2009 Mar 5;360(10):973-84. doi: 10.1056/NEJMoa0808991. PMID 19264686
- [Background] Leckie MJ, ten Brinke A, Khan J, Diamant Z, O'Connor BJ, Walls CM, Mathur AK, Cowley HC, Chung KF, Djukanovic R, Hansel TT, Holgate ST, Sterk PJ, Barnes PJ. Effects of an interleukin-5 blocking monoclonal antibody on eosinophils, airway hyper-responsiveness, and the late asthmatic response. Lancet. 2000 Dec 23-30;356(9248):2144-8. doi: 10.1016/s0140-6736(00)03496-6. PMID 11191542
- [Background] Message SD, Laza-Stanca V, Mallia P, Parker HL, Zhu J, Kebadze T, Contoli M, Sanderson G, Kon OM, Papi A, Jeffery PK, Stanciu LA, Johnston SL. Rhinovirus-induced lower respiratory illness is increased in asthma and related to virus load and Th1/2 cytokine and IL-10 production. Proc Natl Acad Sci U S A. 2008 Sep 9;105(36):13562-7. doi: 10.1073/pnas.0804181105. Epub 2008 Sep 3. PMID 18768794